CLINICAL TRIAL: NCT05123937
Title: Effects of Bobath Technique Versus Task Oriented Training on Gross Motor Function in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LhR/21/0233 Amal Fatima
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOBATH technique (Experimental): In group A (BOBATH) one session per day for three days lasting 1 hour for 3 months. Position transitions such as turning from supine to prone or from prone to supine from sitting to standing are facilitated according to the needs. Balance reflexes are attempted to stimulate by using a CP ball. Ambulation training appropriate to the child's motor development. Additionally, passive stretching of spastic muscle reduces spasticity and facilitates the motor function
  Interventions: Other: BOBATH technique
- Task training (Experimental): In group B (task training) will be applied for 60 minutes per day, 3 times per week for 3 months the individual session lasted roughly 10 minutes for each activity. Standing from a seated situation; (ii) reaching for an object high up, which required ankle plantarflexion from the standing position, and go back to the starting position with the heel leaning on the floor; (iii) stepping on and off a bench; (iv) walking up and downstairs. (10) (v) Drinking water hold the cup stable and drink it by lifting it at an appropriate speed and power (vi) Moving a rubber ball, the task involved taking a 6.5 cm diameter rubber ball and placing it in a basket with a diameter of ten cm (the basket location was moved in various directions).
  Interventions: Other: Task training

INTERVENTIONS:
Other: BOBATH technique — In group A (BOBATH) one session per day for three days lasting 1 hour for 3 months. Position transitions such as turning from supine to prone or from prone to supine from sitting to standing are facilitated according to the needs. Balance reflexes are attempted to stimulate by using a CP ball. Ambulation training appropriate to the child's motor development. Additionally, passive stretching of spastic muscle reduces spasticity and facilitates the motor function
  Arms: BOBATH technique
Other: Task training — In group B (task training) will be applied for 60 minutes per day, 3 times per week for 3 months the individual session lasted roughly 10 minutes for each activity. Standing from a seated situation; (ii) reaching for an object high up, which required ankle plantarflexion from the standing position, and go back to the starting position with the heel leaning on the floor; (iii) stepping on and off a bench; (iv) walking up and downstairs. (10) (v) Drinking water hold the cup stable and drink it by lifting it at an appropriate speed and power (vi) Moving a rubber ball, the task involved taking a 6.5 cm diameter rubber ball and placing it in a basket with a diameter of ten cm (the basket location was moved in various directions).
  Arms: Task training

SUMMARY:
Cerebral palsy is the most familiar motor disorder of childhood. Consistent with the results of recent scientific researches BOBATH approach in physical restoration of youngsters with cerebral palsy promotes formation of motor skills. Improvement in mobility has been primary goal in treatment of CP. There are only a few studies available within the efficacy of "task-oriented training" to improve gross motor function in CP child. Hence, this comparative study is undertaken to gauge the effect of task-oriented training verses neurodevelopmental training on gross motor function in cerebral palsy child. Objective of this study is to find out the effects of BOBATH technique and Task Training on gross motor function in cerebral palsy children. A Convenient sample of Cerebral Palsy children fulfilling inclusion and exclusion criteria, from physiotherapy OPD of Allied & DHQ hospitals of Faisalabad will be considered. Informed consent will be taken from all patient's caregivers. Patients will be divided into two groups through chit draw randomization. Age of children will be 3 years to 10 years without discrimination of gender. Group A will receive BOBATH training and Group B will receive task training. Data will be collected through Gross Motor Function Measure (GMFM-88). Data analyses using SPSS version 25 as a statistical tool.

ELIGIBILITY:
Inclusion Criteria:

Male and female patient Age 3- 10 years. Diagnosed with CP by a specialist. Children with CP GMFCS level I-II. Types of Cerebral palsy (spastic diplegic, quadriplegic, hemiplegic,) without severe abnormalities Cognitive ability should be sufficient that he/she follow simple verbal commands and instructions during training

Exclusion Criteria:

Patient with fixed contracture Patient receiving treatment that affects motor function such as botulinum injection and orthopedic surgery

-

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | Base line and after 3 months
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. The GMFM-88 item scores can be summed to calculate raw and percent scores for each of the five GMFM dimensions of interest selected goal areas and total GMFM-88 scores. The scoring system of the GMFM is a four-point scale divided into five categories (lying and rolling; sitting; crawling and kneeling; standing; walking, running) Reliability refers to dependability, consistency, and stability of scores on an assessment tool. Both versions of GMFM were shown to be highly reliable, with ICCs of greater than .98 (95% confidence interval=0.965-0.994) and both of them can be used in clinical practice or research.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Allied Hospital Faisalabad, Faisalabad, Pakistan(Punjab_, Pakistan

IPD SHARING:
Plan to Share IPD: No